CLINICAL TRIAL: NCT00175318
Title: A Clinical Trial of the Effectiveness of Motivational Interviewing as a Preventive Strategy for Dental Caries in Cree Infants
Brief Title: Testing a Tooth Decay Prevention Program With Cree Mothers and Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Rosamund Harrison, Univerisity of British Columbia
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: B04-0295; PG14R90995
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Dental Caries
Keywords: Motivational interviewing; behavioural modification; maternal counseling
MeSH Terms: conditions — Dental Caries | interventions — Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing — Beginning at 12 months of age, regular application of fluoride varnish will be an option that a mother in the MI group may choose for her child. Control families will receive dental health information from a pamphlet, and will have access to fluoride varnish at local dental clinics.

SUMMARY:
Dental decay is an alarming problem in Cree children. The intervention is a behavioural counseling approach called Motivational Interviewing (MI). The dental health of young children in communities whose mothers had a series of MI sessions provided by Cree women will be compared to the dental health of mothers who did not have the intervention.

DETAILED DESCRIPTION:
Dental decay is an alarming problem in Cree children. The intervention is a behavioural counseling approach called Motivational Interviewing (MI). The dental health of young children in communities whose mothers had a series of MI sessions provided by Cree women will be compared to the dental health of mothers who did not have the intervention.

The proposed randomized controlled trial, involving Cree mothers and children in Eeyou Istchee, will test the effectiveness of an innovative, one-on-one counseling program called Motivational Interviewing (MI). In keeping with Cree philosophy and traditions, MI allows mothers to choose from a "menu" of preventive dental behaviours. The primary research question is whether there will be any difference in the dental health status of Cree children from communities where mothers have participated in MI interventions, compared to children from communities where mothers received information by more traditional means (pamphlets). This question will be answered by testing the hypothesis that the prevalence of caries among children 30 months of age will be lower in experimental "MI" communities than in control communities. The secondary questions are whether Cree mothers' beliefs about child dental health, children's dental health practices, and the negative health outcomes of ECC will be altered in MI communities compared to control communities.

Trial design: Over the past two years, the project team has undertaken extensive community consultation to better understand the problem of dental caries in young Cree children, and to seek community input for the project. The design is single blind, with cluster randomization by community, and two treatment groups. A total study sample of 309 mother-child pairs accounts for attrition of 15% over 3 years, and for infant mortality. The power is 82% to detect a 20% reduction in caries prevalence. The "experimental" treatment, MI, will assist mothers to choose from a menu of various age-appropriate, preventive options. The first intervention will occur during pregnancy, followed by regular MI sessions beginning at the child's 2-month immunization until 24 months of age. Local Cree dental assistants, following training and calibration in the MI technique, will do the counseling. Beginning at 12 months of age, regular application of fluoride varnish will be an option that a mother in the MI group may choose for her child. Control families will receive dental health information from a pamphlet, and will have access to fluoride varnish at local dental clinics.

Outcomes assessment: To answer the first research question, calibrated dentists from outside of Eeyou Istchee will do dental examinations for children at 30+3 months of age. Mothers will complete questionnaires to answer the secondary questions. The primary statistical analysis will be a comparison of caries prevalence in intervention and control groups, using a permutation test with test statistic equal to the difference between caries prevalences in the two groups. A significance level will be determined using the exact permutation distribution of the test statistic, which will be computed by enumerating all possible random assignments of villages to intervention or control conditions according to the randomization scheme..

ELIGIBILITY:
Inclusion Criteria:

First Nations women from the 9 communities of Eeyou Istchee (Cree territory of James Bay, Quebec) who are pregnant or have a pre-dentate infant l

Exclusion Criteria:

Ages: 14 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 309 (Estimated)
Dates: Start 2005-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Dental health status of children 30 months of age in test and control communities | 24 months

SECONDARY OUTCOMES:
Mothers' beliefs about child dental health, children's dental health practices, and the negative health outcomes of dental caries assessed at project's end. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Rosamund Harrison, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Cree Board of Health and Social Services of James Bay, Chisasibi, Quebec, Canada

REFERENCES:
- [Result] Harrison R, Veronneau J, Leroux B. Design and implementation of a dental caries prevention trial in remote Canadian Aboriginal communities. Trials. 2010 May 13;11:54. doi: 10.1186/1745-6215-11-54. PMID 20465831